CLINICAL TRIAL: NCT02431208
Title: A Phase Ib Study of the Safety and Pharmacokinetics of Atezolizumab (Anti-PD-L1 Antibody) Alone or in Combination With an Immunomodulatory Drug and/or Daratumumab in Patients With Multiple Myeloma (Relapsed/Refractory and Post-Autologous Stem Cell Transplantation)
Brief Title: A Study of Atezolizumab (Anti-Programmed Death-Ligand 1 [PD-L1] Antibody) Alone or in Combination With an Immunomodulatory Drug and/or Daratumumab in Participants With Multiple Myeloma (MM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29695
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — atezolizumab; Atazanavir Sulfate; daratumumab; Lenalidomide; pomalidomide; Dexamethasone

ARMS (11):
- Cohort A: ATZ (Run-In) (Experimental): Cohort A will involve a safety run-in to evaluate atezolizumab administered as a single agent in participants with relapsed or refractory MM who have received up to 3 lines of prior treatment. NOTE: This cohort has been completed.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody
- Cohort B1: ATZ + LEN (Dose Escalation) (Experimental): Cohort B1 will involve a dose escalation to evaluate atezolizumab administered in combination with ascending-dose lenalidomide in participants with relapsed or refractory MM who have received up to 3 lines of prior treatment. NOTE: This cohort has been completed.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody; Drug: Lenalidomide
- Cohort C: ATZ + LEN (Post-ASCT): (Experimental): Cohort C will evaluate atezolizumab administered in combination with lenalidomide in participants with MM who have measureable disease after ASCT. NOTE: This cohort is closed to enrollment.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody; Drug: Lenalidomide
- Cohort D1: ATZ + DAR (Run-in) (Experimental): Cohort D1 will involve a safety run-in to evaluate atezolizumab administered in combination with daratumumab in participants with relapsed or refractory MM who have received up to 3 lines of prior treatment.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody; Drug: Daratumumab
- Cohort D2: ATZ + DAR (Expansion) (Experimental): Cohort D2 will involve an expansion to evaluate atezolizumab administered in combination with daratumumab in participants with relapsed or refractory MM who have received 2 but no more than 3 lines of prior treatment that must have included a PI and IMiD and are refractory to the last line of treatment.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody; Drug: Daratumumab
- Cohort D3: ATZ + DAR (Progressed) (Experimental): Cohort D3 will involve an expansion to evaluate atezolizumab in combination with daratumumab in participants with relapsed or refractory MM who have received 2 or more lines of prior treatment and have progressed with an anti-cluster of differentiation (CD) 38 monoclonal antibody, either alone or in combination, and are refractory to both a proteasome inhibitor (PI) and immunomodulatory drug (IMiD).
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody; Drug: Daratumumab
- Cohort E1: ATZ + DAR + LEN (Dose Escalation) (Experimental): Cohort E1 will involve a dose escalation to evaluate atezolizumab administered in combination with daratumumab and ascending-dose lenalidomide in participants with relapsed or refractory MM who have received up to 3 lines of prior treatment. NOTE: This cohort is closed to enrollment.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody; Drug: Daratumumab; Drug: Lenalidomide
- Cohort E2: ATZ + DAR + LEN (Expansion) (Experimental): Cohort E2 will involve an expansion to evaluate atezolizumab administered in combination with daratumumab and the maximum tolerated dose (MTD) of lenalidomide determined in Cohort E1 in participants with relapsed or refractory MM who have received up to 3 lines of prior treatment. NOTE: This cohort is closed to enrollment.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody; Drug: Daratumumab; Drug: Lenalidomide
- Cohort F1: ATZ + DAR + POM (Dose Escalation) (Experimental): Cohort F1 will involve a dose escalation to evaluate atezolizumab administered in combination with daratumumab and ascending-dose pomalidomide in participants with relapsed or refractory MM who have received 4 or more lines of prior treatment and are refractory to the last line of treatment. NOTE: This cohort has been completed.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody; Drug: Daratumumab; Drug: Pomalidomide
- Cohort F2: ATZ + DAR + POM (Expansion) (Active Comparator): Cohort F2 will involve an expansion to evaluate atezolizumab administered in combination with daratumumab and the MTD of pomalidomide determined in Cohort F1 in participants with relapsed or refractory MM who have received 4 or more lines of prior treatment and are refractory to the last line of treatment. NOTE: This cohort is randomized.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody; Drug: Daratumumab; Drug: Pomalidomide
- Cohort F3: DAR + POM + Dexamethasone (Active Comparator): Cohort F3 is an expansion control arm for cohort F2. Participants will receive daratumumab in combination with pomalidomide at the MTD and dexamethasone. NOTE: This cohort is randomized.
  Interventions: Drug: Daratumumab; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody — Participants will receive intravenous (IV) atezolizumab until loss of clinical benefit, withdrawal, or study end. Cohorts A to C will receive 1200 milligrams (mg) on Day 1 of each 21-day cycle. Cohorts D to F (combination with daratumumab) will receive 840 mg on Days 2 and 16 of Cycle 1 and on Days 1 and 15 of each 28-day cycle thereafter.
  Other Names: Tecentriq, MPDL3280A, "ATZ"
  Arms: Cohort A: ATZ (Run-In); Cohort B1: ATZ + LEN (Dose Escalation); Cohort C: ATZ + LEN (Post-ASCT):; Cohort D1: ATZ + DAR (Run-in); Cohort D2: ATZ + DAR (Expansion); Cohort D3: ATZ + DAR (Progressed); Cohort E1: ATZ + DAR + LEN (Dose Escalation); Cohort E2: ATZ + DAR + LEN (Expansion); Cohort F1: ATZ + DAR + POM (Dose Escalation); Cohort F2: ATZ + DAR + POM (Expansion)
Drug: Daratumumab — Participants will receive 16 milligrams per kilogram (mg/kg) IV daratumumab until loss of clinical benefit, withdrawal, or study end. Treatment will be per the U.S. Package Insert and given on Days 1, 8, 15, 22 of Cycles 1 and 2; on Days 1 and 15 of Cycles 3 to 6; and on Day 1 of each 28-day cycle thereafter.
  Other Names: Darzalex, "DAR"
  Arms: Cohort D1: ATZ + DAR (Run-in); Cohort D2: ATZ + DAR (Expansion); Cohort D3: ATZ + DAR (Progressed); Cohort E1: ATZ + DAR + LEN (Dose Escalation); Cohort E2: ATZ + DAR + LEN (Expansion); Cohort F1: ATZ + DAR + POM (Dose Escalation); Cohort F2: ATZ + DAR + POM (Expansion); Cohort F3: DAR + POM + Dexamethasone
Drug: Lenalidomide — Lenalidomide will be administered orally (PO) until loss of clinical benefit, withdrawal, or study end. Cohort B1 will receive 10, 15, or 25 mg, ascending-dose lenalidomide, on Days 1-14 of each 21-day cycle. Cohort C will receive 10 mg on Days 1-14 of each 21-day cycle, beginning in Cycle 4. Cohort E (combination with daratumumab) will receive 10, 15, or 25 mg on Days 1-21 of each 28-day cycle. Participants in Cohort E1 will receive ascending-dose lenalidomide, and those in Cohort E2 will receive lenalidomide at the MTD as determined in Cohort E1.
  Other Names: Revlimid, "LEN"
  Arms: Cohort B1: ATZ + LEN (Dose Escalation); Cohort C: ATZ + LEN (Post-ASCT):; Cohort E1: ATZ + DAR + LEN (Dose Escalation); Cohort E2: ATZ + DAR + LEN (Expansion)
Drug: Pomalidomide — Pomalidomide will be administered PO until loss of clinical benefit, withdrawal, or study end. Cohort F (combination with daratumumab) will receive 2 or 4 mg on Days 1-21 of each 28-day cycle. Participants in Cohort F1 will receive ascending-dose pomalidomide, and those in Cohort F2 will receive pomalidomide at the MTD as determined in Cohort F1.
  Other Names: Pomalyst, "POM"
  Arms: Cohort F1: ATZ + DAR + POM (Dose Escalation); Cohort F2: ATZ + DAR + POM (Expansion); Cohort F3: DAR + POM + Dexamethasone
Drug: Dexamethasone — Participants will receive either 20mg or 40mg of dexamethasone PO every 7 days from Day 1 of each cycle.
  Arms: Cohort F3: DAR + POM + Dexamethasone

SUMMARY:
This multicenter, open-label, Phase I study will evaluate the safety, efficacy, and pharmacokinetics of atezolizumab alone or in combination with daratumumab and/or various immunomodulatory agents in participants with MM who have relapsed or who have undergone autologous stem cell transplantation (ASCT). Cycle length will be 21 days in Cohorts A to C and 28 days in Cohorts D to F.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of MM with objective evidence of measurable disease
* Willing and able to undergo bone marrow aspiration and biopsy tissue sample collection during screening and on study
* Eastern Cooperative Oncology Group (ECOG) performance status score less than or equal to (</=) 2
* Left ventricular ejection fraction (LVEF) greater than or equal to (>/=) 40 percent (%)
* Total bilirubin </=2 times the ULN
* Creatinine </=2.0 milligrams per deciliter (mg/dL), with creatinine clearance (CrCl) using the Cockcroft-Gault formula >/=40 milliliters per minute (mL/min) or 60 mL/min for those who receive lenalidomide
* Corrected calcium at or below ULN
* Transaminase levels </=2.5 times the upper limit of normal (ULN)
* Receipt of >/=1 but not more than 3 prior lines of therapy (Cohorts A, B, C, D1, E)
* Receipt of 2, but not more that 3 prior lines of therapy that must have included a proteasome inhibitor (PI) and immunomodulatory drug (IMiD) (alone or in combination, and are refractory to the last line of treatment(Cohort D2)
* Receipt of >/=2 prior lines of therapy and progressed on treatment with an anti-CD38 monoclonal antibody and are refractory to both a PI and IMiD (Cohort D3)
* Receipt of >/=4 lines of prior therapy and are refractory to the last line of treatment (Cohort F)
* Absolute neutrophil count (ANC) >/=1000 cells per microliter (cells/mcL) (Cohorts A, B, D, E, F)
* Platelet count >/=50,000 cells/mcL, or >/=30,000 cells/mcL if more than 50% bone marrow involvement (Cohorts A, B, D, E, F)
* All participants who are prescribed lenalidomide or pomalidomide must be counseled at a minimum of every 21-28 days about pregnancy precautions and risks of fetal exposure (Cohorts B, C, E, F)
* Agree to be registered in and comply with all requirements of the Revlimid Risk Evaluation and Mitigation Strategy (REMS) program (Cohorts B, C, E)
* Agree to be registered in and comply with all requirements of the Pomalyst REMS program (Cohort F)
* Sufficient recovery from first or second ASCT within 60-120 days of transplant (Cohort C)
* Off antibiotic/antifungal therapy for >/=14 days (Cohort C)
* Completion of any prior radiotherapy (Cohort C)
* ANC >/=1500 cells/mcL (Cohort C)

Exclusion Criteria:

* Other malignancy within 2 years prior to screening, with some exceptions
* Prior therapy with atezolizumab or other immunotherapies including CD137 agonists, anti-programmed death (PD)-1, anti-cytotoxic T-lymphocyte associated protein 4 (CTLA-4), and anti-PD-L1 therapeutic antibodies
* Uncontrolled cancer pain
* Treatment with any investigational drug within 30 days or 5 half-lives of the investigational drug, whichever is longer
* Known hypersensitivity to study drug and/or drug class
* History of autoimmune disease except for controlled, treated thyroidism or Type 1 diabetes
* Prior systemic anti-myeloma therapy within 14 days of Cycle 1 Day 1
* Prior treatment with chimeric antigen receptor (CAR) T cells or other forms of adoptive cellular therapy, with the exception of autologous stem cell transplantation
* Polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes (POEMS) syndrome
* Plasma cell leukemia (greater than 2,000 cells/mcL of circulating plasma cells by standard differential)
* Immunosuppressive therapy within 6 weeks of Cycle 1 Day 1
* Daily corticosteroid requirement within 2 weeks of Cycle 1 Day 1
* Prior allogeneic stem cell transplant or solid organ transplant
* Active hepatitis B, active hepatitis C, or positive for human immunodeficiency virus (HIV)
* Uncontrolled, clinically significant pulmonary disease (for example, chronic obstructive pulmonary disease, pulmonary hypertension, idiopathic pulmonary fibrosis) that in the opinion of the investigator would put the participant at significant risk for pulmonary complications during the study
* History of pneumonitis
* Uncontrolled intercurrent illness including but not limited to uncontrolled infection, disseminated intravascular coagulation, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding females
* Inability to tolerate thromboprophylaxis (Cohorts B, C, E, F)
* Evidence of progressive MM compared to pretransplant evaluation (Cohort C)
* Prior treatment with anti-CD38 therapy including daratumumab (Cohorts D1, D2, E, F)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants by Best Overall Response According to International Myeloma Working Group (IMWG) Criteria | From Day 1 of Cycle 2 (cycle = 21 or 28 days) until progression, withdrawal, or study end (up to 36 months overall)
Recommended Phase II Dose (RP2D) of Lenalidomide in the Combinations Tested | From start of treatment until 30 days after last dose (up to approximately 36 months)
RP2D of Pomalidomide in the Combinations Tested | From start of treatment until 30 days after last dose (up to approximately 36 months)
Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | From start of treatment until 30 days after last dose (up to approximately 36 months)

SECONDARY OUTCOMES:
Duration of Response (DOR) According to IMWG Criteria | From first observed response until the date of first recorded progression or death from any cause (up to 36 months overall)
Progression-Free Survival (PFS) According to IMWG Criteria | From start of treatment until the date of first recorded progression or death from any cause (up to 36 months overall)
Percentage of Participants with Objective Response According to IMWG Criteria | From Day 1 of Cycle 2 until progression, withdrawal, or study end (up to 36 months overall). For Cohort D3 Only: 6, 9, and 12 months.
Overall Survival | From start of treatment until death from any cause (up to 36 months overall)
Maximum Observed Serum Concentration (Cmax) of Atezolizumab | From predose (0 hours [h]) on Day 1 of Cycle 1 until treatment discontinuation (up to 36 months overall); see Outcome Measure Description for details
  Predose (0 h) and postdose (0.5 h) (infusion = 0.5-1 h) on Day 1 of Cycles 1, 3 (cycle = 21 or 28 days) and Day 2 of Cycle 1; predose (0 h) on Day 1 of Cycles 2, 4, 8; then every 8 cycles until/at treatment discontinuation (up to 36 months); and 90 days after last dose (up to 36 months overall)
Minimum Observed Serum Concentration (Cmin) of Atezolizumab | Predose (0 h) on Day 1 of Cycles 1, 2, 3, 4, 8 (cycle = 21 or 28 days) and Day 2 of Cycle 1; then every 8 cycles until/at treatment discontinuation (up to 36 months); and 90 days after last dose (up to 36 months overall)
Cmax of Lenalidomide | Predose (0 h) and postdose (1 h) on Day 1 of Cycles 1, 4 (cycle = 21 days); predose (0 h) and postdose (0.5, 1, 2, 4, 8 h) on Day 15 of Cycles 1, 3; predose (0 h) and postdose (2 h) on Day 15 of Cycles 2, 4, 8
Cmin of Lenalidomide | Predose (0 h) on Day 1 of Cycles 1, 4 (cycle = 21 days) and Day 15 of Cycles 1, 2, 3, 4, 8
Cmax of Pomalidomide | Predose (0 h) and postdose (1, 2, 4, 6, 8 h) on Day 15 of Cycles 1, 3 (cycle = 28 days); predose (0 h) and postdose (4 h) on Day 15 of Cycles 2, 4, 8
Cmin of Pomalidomide | Predose (0 h) on Day 15 of Cycles 1, 2, 3, 4, 8 (cycle = 28 days)
Cmax of Daratumumab | From predose (0 h) on Day 1 of Cycle 1 until treatment discontinuation (up to 36 months overall); see Outcome Measure Description for details
  Predose (0 h) and postdose (0.5 h) (infusion ~3-6 h) on Day 1 of Cycles 1, 3 (cycle = 28 days); predose (0 h) on Day 1 of Cycles 2, 4, 8; then every 8 cycles until/at treatment discontinuation (up to 36 months); and 90 days after last dose (up to 36 months overall)
Cmin of Daratumumab | Predose (0 h) on Day 1 of Cycles 1, 2, 3, 4, 8 (cycle = 28 days); then every 8 cycles until/at treatment discontinuation (up to 36 months); and 90 days after last dose (up to 36 months overall)
Change in Number of Participants With Anti-Drug Antibody (ADA) Response to Atezolizumab from Baseline to End of Study | From treatment start until study end (up to 36 months overall); see Outcome Measure Description for details
  From treatment start until study end; assessed predose (0 h) on Day 1 of Cycles 1, 2, 3, 4, 8 (cycle = 21 or 28 days) and Day 2 of Cycle 1; then every 8 cycles until/at treatment discontinuation (up to 36 months); and 90 days after last dose (up to 36 months overall)
Change in Number of Participants With ADA Response to Daratumumab from Baseline to End of Study | From treatment start until study end; assessed predose (0 h) on Day 1 of Cycles 1, 3, 8 (cycle = 28 days); at treatment discontinuation (up to 36 months); and 90 days after last dose (up to 36 months overall)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (31):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University Of Arkansas, Little Rock, Arkansas
  - Scripps Clinic Torrey Pines, La Jolla, California
  - UC Davis; Comprehensive Cancer Center, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Mayo Clinic Hospital - Florida, Jacksonville, Florida
  - Emory Univ Winship Cancer Inst, Atlanta, Georgia
  - Loyola University Med Center, Maywood, Illinois
  - Indiana University Health; Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University Department of Medicine; IU Simon Cancer Center, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr; Hem/Onc, Boston, Massachusetts
  - Univ of Michigan Medical Ctr, Ann Arbor, Michigan
  - Karmanos Cancer Institute., Detroit, Michigan
  - Henry Ford Hospital; Hematology Oncology, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Mount SInai Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center; Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Lifespan Cancer Institute, Providence, Rhode Island
  - Medical University of South Carolina; Hollings Cancer Center, Charleston, South Carolina
  - Texas Oncology-Baylor Sammons Cancer Center, Dallas, Texas
  - UT Southwestern MC at Dallas, Dallas, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Derived] Wong S, Hamidi H, Costa LJ, Bekri S, Neparidze N, Vij R, Nielsen TG, Raval A, Sareen R, Wassner-Fritsch E, Cho HJ. Multi-omic analysis of the tumor microenvironment shows clinical correlations in Ph1 study of atezolizumab +/- SoC in MM. Front Immunol. 2023 Jul 25;14:1085893. doi: 10.3389/fimmu.2023.1085893. eCollection 2023. PMID 37559718